CLINICAL TRIAL: NCT00357370
Title: A Pilot Study of the Efficacy and Safety of BMS-512148 on Glycemic Control in Subjects With Type 2 Diabetes Treated Aggressively But Not Controlled on Combination Antihyperglycemic Therapy With Metformin and/or Thiazolidinedione (TZD) and Insulin.
Brief Title: A Pilot Study of BMS-512148 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB102-009
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 20 mg
  Interventions: Drug: Dapagliflozin
- Cohort 2 - Arm 1 (Experimental): 10 mg
  Interventions: Drug: Dapagliflozin
- Cohort 2 - Arm 2 (Experimental): 20 mg
  Interventions: Drug: Dapagliflozin
- Cohort 2 - Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, once daily, up to 12 weeks
  Other Names: BMS-512148
  Arms: Cohort 1; Cohort 2 - Arm 1; Cohort 2 - Arm 2
Drug: Placebo — Tablets, Oral, 0 mg, once daily, up to 12 weeks
  Arms: Cohort 2 - Arm 3

SUMMARY:
The purpose of this clinical research study is to learn if BMS-512148, added to insulin and one or two anti-diabetes medications (metformin and/or pioglitazone or rosiglitazone), can help reduce the blood sugar levels compared to insulin and one or two anti-diabetes medications (metformin and/or pioglitazone or rosiglitazone) alone, in subjects with type 2 diabetes. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 to 75 years old, with type 2 diabetes with inadequate glycemic control
* Subjects receiving insulin and metformin and/or a thiazolidinedione
* Body Mass Index <=45.0 kg/m2
* Serum creatinine <1.5 mg/dL for men or <1.4 mg/dL for women
* No overt proteinuria (in subjects with a microalbumin/creatinine ratio ≥300 mg/g, the 24-hour urinary excretion of total protein must be <3 g/24 hrs)

Exclusion Criteria:

* History of type 1 diabetes
* AST and/or ALT >2.5 times the upper limit of normal
* Creatinine kinase ≥3 times the upper limit of normal
* Symptoms of severely uncontrolled diabetes
* History of hypoglycemic unawareness
* Currently unstable or serious cardiovascular, renal, hepatic, hematological, oncological, endocrine, psychiatric, or rheumatic diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2006-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (23):
- United States (16):
  - Nea Clinic, Jonesboro, Arkansas
  - Valley Research, Fresno, California
  - Bernstein, Richard, Greenbrae, California
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Indiana University, Indianapolis, Indiana
  - Model Clinical Research Llc, Baltimore, Maryland
  - University Of Michigan, Ann Arbor, Michigan
  - St. Louis Center For Clinical Research, St Louis, Missouri
  - Suny Upstate Medical University, Syracuse, New York
  - Mountain Diabetes And Endocrine Center, Asheville, North Carolina
  - Your Diabetes Endocrine Nutrition Group, Mentor, Ohio
  - Research Institute Of Dallas, P.A., Dallas, Texas
  - Diabetes And Glandular Disease Research Associates, P.A., San Antonio, Texas
  - Rainier Clinical Research Center, Renton, Washington
  - Advanced Healthcare S.C., Milwaukee, Wisconsin
- Canada (7):
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Bathurst, New Brunswick
  - Local Institution, Gatineau, Quebec
  - Local Institution, Laval, Quebec
  - Local Institution, Longueuil, Quebec
  - Local Institution, Pointe-Claire, Quebec
  - Local Institution, Sherbrooke, Quebec

REFERENCES:
- [Result] Wilding JP, Norwood P, T'joen C, Bastien A, List JF, Fiedorek FT. A study of dapagliflozin in patients with type 2 diabetes receiving high doses of insulin plus insulin sensitizers: applicability of a novel insulin-independent treatment. Diabetes Care. 2009 Sep;32(9):1656-62. doi: 10.2337/dc09-0517. Epub 2009 Jun 15. PMID 19528367
- [Derived] Mellander A, Billger M, Johnsson E, Traff AK, Yoshida S, Johnsson K. Hypersensitivity Events, Including Potentially Hypersensitivity-Related Skin Events, with Dapagliflozin in Patients with Type 2 Diabetes Mellitus: A Pooled Analysis. Clin Drug Investig. 2016 Nov;36(11):925-933. doi: 10.1007/s40261-016-0438-3. PMID 27461213
- [Derived] Kohan DE, Fioretto P, Johnsson K, Parikh S, Ptaszynska A, Ying L. The effect of dapagliflozin on renal function in patients with type 2 diabetes. J Nephrol. 2016 Jun;29(3):391-400. doi: 10.1007/s40620-016-0261-1. Epub 2016 Feb 19. PMID 26894924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 163 participants enrolled, Of these 163 participants, 71 were randomized and received treatment. Of these 71 participants, 60 completed double-blind treatment period
Groups:
- Dapagliflozin 20 mg; Placebo; Dapagliflozin 10 mg: Tablets, oral, once daily for 12 weeks
Period: Cohort 1
Arm/Group | Dapagliflozin 20 mg | Placebo | Dapagliflozin 10 mg
Started | 4 | 0 | 0
Completed | 4 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Cohort 2
Arm/Group | Dapagliflozin 20 mg | Placebo | Dapagliflozin 10 mg
Started | 24 | 23 | 24
Completed | 22 | 16 | 22
Not Completed | 2 | 7 | 2
Not completed — Lack of Efficacy | 0 | 2 | 1
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — non-compliance, not met criteria, etc | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients who received at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 20 mg | Placebo | Dapagliflozin 10 mg | Total
Number analyzed (Participants) | 24 | 23 | 24 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.1 (10.63) | 58.4 (6.49) | 55.7 (9.20) | 56.7 (8.92)
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 20 | 19 | 20 | 59
  65 years or older | 4 | 4 | 4 | 12
Sex/Gender, Customized [Number; unit: Participants]
  Male | 13 | 16 | 13 | 42
  Female | 11 | 7 | 11 | 29
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 23 | 22 | 22 | 67
  Back/African American | 1 | 0 | 1 | 2
  Asian | 0 | 0 | 1 | 1
  Other | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1C (HbA1c) at Week 12 (Last Observation Carried Forward [LOCF]) - Cohort 2
Description: HbA1c was measured as percent of hemoglobin by a central laboratory. Data after insulin uptitration was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. HbA1c measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 4, 6, 8, 10, and 12 in the double-blind period.
Time Frame: From Baseline to Week 12
Population: Chort 2 all randomized participants who received study medication and had nonmissing HbA1c values at baseline and Week 12 (LOCF). Note: participants in cohort 1 provided data to establish an acceptable safety and tolerability profile when dapagliflozin 20 mg was added to open-label oral antidiabetic agent plus insulin.
Measure: Mean (Standard Error); unit: % of hemoglobin
Arm/Group | Placebo | Dapagliflozin 10 mg | Dapagliflozin 20 mg
Number analyzed (Participants) | 19 | 23 | 23
% of hemoglobin | 0.09 (0.1406) | -0.61 (0.1276) | -0.69 (0.1278)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.08 to -0.32], Standard Error of Mean 0.1898 — ANCOVA was applied. No formal statistical testing was performed to compare between treatment groups
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 20 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.16 to -0.40], Standard Error of Mean 0.1903 — ANCOVA was applied. No formal statistical testing was performed to compare between treatment groups

2. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 12 (Last Observation Carried Forward [LOCF]) - Cohort 2
Description: Fasting plasma glucose was measured as milligrams per deciliter(mg/dL) by a central laboratory. Data after insulin uptitration was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. FPG measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 1, 2, 4, 6, 8, 10, and 12 in the double-blind period.
Time Frame: From Baseline to Week 12
Population: Chort 2 all randomized participants who received study medication and had nonmissing FPG values at baseline and Week 12 (LOCF). Note: participants in cohort 1 provided data to establish an acceptable safety and tolerability profile when dapagliflozin 20 mg was added to open-label oral antidiabetic agent plus insulin.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Dapagliflozin 10 mg | Dapagliflozin 20 mg
Number analyzed (Participants) | 22 | 23 | 23
mg/dL | 17.80 (8.1941) | 2.36 (7.9992) | -9.64 (7.9908)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -15.44, 95% CI 2-sided [-38.37 to 7.48], Standard Error of Mean 11.4753 — ANCOVA was applied. No formal statistical testing was performed to compare between treatment groups
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 20 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -27.44, 95% CI 2-sided [-50.33 to -4.55], Standard Error of Mean 11.4574 — ANCOVA was applied. No formal statistical testing was performed to compare between treatment groups

3. Secondary Outcome: Participants Achieving a Therapeutic Glycemic Response (Hemoglobin A1c [HbA1C]) <7.0% at Week 12 (Last Observation Carried Forward [LOCF]) - Cohort 2
Description: Therapeutic glycemic response is defined as HbA1c <7.0%. Data after insulin uptitration was excluded from this analysis. HbA1c was measured as a percent of hemoglobin.
Time Frame: From Baseline to Week 12
Population: Chort 2 all randomized participants who received study medication and had nonmissing values at baseline and Week 12 (LOCF). Note: participants in cohort 1 provided data to establish an acceptable safety and tolerability profile when dapagliflozin 20 mg was added to open-label oral antidiabetic agent plus insulin.
Measure: Number; unit: Participants
Arm/Group | Placebo | Dapagliflozin 10 mg | Dapagliflozin 20 mg
Number analyzed (Participants) | 19 | 23 | 23
Participants | 1 (5.3) | 3 (13.0) | 1 (4.3)

4. Secondary Outcome: Participants Achieving a Therapeutic Glycemic Response (Hemoglobin A1c [HbA1C]) <=6.5% at Week 12 (Last Observation Carried Forward [LOCF]) - Cohort 2
Description: Therapeutic glycemic response is defined as HbA1c <=6.5%. Data after insulin uptitration was excluded from this analysis. HbA1c was measured as a percent of hemoglobin.
Time Frame: From Baseline to Week 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Dapagliflozin 10 mg | Dapagliflozin 20 mg
Number analyzed (Participants) | 19 | 23 | 23
Participants | 0 (5.3) | 1 (13.0) | 0 (4.3)

5. Secondary Outcome: Participants Achieving a Therapeutic Glycemic Response (Hemoglobin A1c [HbA1C]) Decrease From Baseline >= 0.5% at Week 12 (Last Observation Carried Forward [LOCF]) - Cohort 2
Description: Therapeutic glycemic response is defined as HbA1c decrease from baseline >= 0.5% at Week 12. Data after insulin uptitration was excluded from this analysis. HbA1c was measured as a percent of hemoglobin.
Time Frame: From Baseline to Week 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Dapagliflozin 10 mg | Dapagliflozin 20 mg
Number analyzed (Participants) | 19 | 23 | 23
Participants | 3 (5.3) | 15 (13.0) | 15 (4.3)

6. Secondary Outcome: Adjusted Mean Total Daily Dose of Insulin (TDDI) Change From Baseline at Week 12 (LOCF), Including Data After Up-titration of Insulin) - Cohort 2
Description: Baseline TDDI was reduced by 50% prior to treatment, except 2 subjects. TDDI could be up-titrated according to prespecified criteria at Weeks 4, 6, 8, 10 and 12 in the double-blind period.
Time Frame: From Baseline to Week 12
Population: Chort 2 all randomized participants who received study medication and had nonmissing TDDI values at baseline and Week 12 (LOCF). Note: participants in cohort 1 provided data to establish an acceptable safety and tolerability profile when dapagliflozin 20 mg was added to open-label oral antidiabetic agent plus insulin.
Measure: Mean (Standard Error); unit: units/day
Arm/Group | Placebo | Dapagliflozin 10 mg | Dapagliflozin 20 mg
Number analyzed (Participants) | 22 | 24 | 24
units/day | 1.69 (2.7659) | -1.35 (2.6489) | -0.83 (2.6484)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 10 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -3.05, 95% CI 2-sided [-10.69 to 4.60], Standard Error of Mean 3.8302 — ANCOVA was applied. No formal statistical testing was performed to compare between treatment groups
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 20 mg; Test type: Superiority or Other; Mean Difference (Final Values) = -2.52, 95% CI 2-sided [-10.17 to 5.12], Standard Error of Mean 3.8291 — ANCOVA was applied. No formal statistical testing was performed to compare between treatment groups

ADVERSE EVENTS:
Time Frame: Onset on or after the first date of double-blind treatment and on or prior to the last day of double-blind treatment 12 weeks plus 4 days for non-serious adverse event; plus 30 days for serious adverse event.
Arm/Group | Dapagliflozin 20 mg | Placebo | Dapagliflozin 10 mg
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/23 | 0/24
Other Adverse Events (participants affected / at risk) | 13/24 | 12/23 | 12/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 20 mg (N=24) | Placebo (N=23) | Dapagliflozin 10 mg (N=24)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 20 mg (N=24) | Placebo (N=23) | Dapagliflozin 10 mg (N=24)
NAUSEA (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (3)
POLLAKIURIA (Renal and urinary disorders) | 3 (3) | 4 (5) | 2 (3)
VOMITING (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3)
DRY MOUTH (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 2 (6) | 2 (2) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 2 (2)
INFLUENZA (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
THIRST (General disorders) | 1 (1) | 1 (1) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (2) | 2 (4) | 2 (4)
HEADACHE (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Cohort 1 data provided information on insulin dose adjustment (n=4).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No